CLINICAL TRIAL: NCT03561233
Title: Prevalence and Predictors of Proton Pump Inhibitor Partial Response in Gastroesophageal Reflux Disease in Systemic Sclerosis
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Khon Kaen University (Other)
Collaborators: Thai Rheumatism Association (Unknown)
Responsible Party: Principal Investigator, Chingching Foocharoen, Principle investigator, Khon Kaen University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PPI partial response GERD SSc
Record Dates: First submitted 2018-06-07; First posted 2018-06-19 (Actual); Last update posted 2018-06-21 (Actual); Status verified 2018-06

CONDITIONS: Systemic Sclerosis; Gastroesophageal Reflux; Proton Pubm Inhibitor
MeSH Terms: conditions — Scleroderma, Systemic; Gastroesophageal Reflux | interventions — Omeprazole

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- proton pump inhibitor (Experimental): omeprazole 20 mg twice daily
  Interventions: Drug: Omeprazole 20mg

INTERVENTIONS:
Drug: Omeprazole 20mg — omeprazole 20 mg twice daily 30 minutes before meal for 4 weeks

SUMMARY:
Proton pump inhibitor (PPI) twice daily dosing regimen-a standard dose therapy for gastroesophageal reflux disease (GERD)-is an effective therapy for uncomplicated GERD in systemic sclerosis (SSc) but there is no data of response rate of standard dose of PPI and predictors of PPI-partial response (PPI-PR) GERD in SSc.Objectives of the study were to determine the prevalence of omeprazole partial response GERD in SSc and to define the predictors of PPI-PR GERD in SSc. Adult SSc patients having GERD were treated with omeprazole 20 mg twice daily 30 minutes before meal for 4 weeks. Severity of symptom-grading by visual analogue scale (VAS) and frequency of symptoms by frequency scale for symptoms of GERD (FSSG) were assessed at baseline and 4 weeks after treatment. PPI-PR GERD was defined by less than 50% improvement in VAS of severity of symptom and acid reflux score by FSSG after treatment compare to baseline.

ELIGIBILITY:
Inclusion Criteria:

1. SSc patients aged between 18 and 65 years.
2. Clinically diagnosed as GERD
3. Must not receive any PPI or prokinetic drug within 2 weeks before baseline evaluation

Exclusion Criteria:

1. Pregnancy or lactation
2. Previous history of gastroesophageal surgery or endoscopic therapy due to severe erosive esophagitis
3. Present of Barrett's esophagus
4. Bedridden and confined to no self-care
5. Evidence of active malignant disease
6. Present of uncontrolled or severe medical problems such as asthma, angina, hepatic or renal diseases
7. Present of active infection that needs systemic antibiotic
8. Allergic history of omeprazole
9. Receiving prohibit co-medications that may have drug interaction or attenuate GERD symptoms such as tetracycline, ferrous salt, digoxin, isoniacid, oral bisphosphonate

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 250 (Actual)
Dates: Start 2013-05 (Actual); Primary Completion 2018-05 (Actual); Study Completion 2018-06 (Actual)

PRIMARY OUTCOMES:
Changing severity of heart burn of SSc related GERD evaluated by visual analogue score (VAS) Changing Severity of Heart Burn of SSc Evaluated by Visual Analogue Score (VAS) | 4 weeks
  VAS scale 0-100 was applied for an outcome measurement of the severity of heart burn. The VAS scale 0 was no symptoms of heart burn and scale 100 was a maximum symptom of heart burn. The changing of the severity of heart burn was the changing of VAS before and after treatment. PPI-PR GERD is defined when the changing of severity of heart burn is improvement less than 50% compare to baseline.
Changing of Frequency of Symptoms in SSc related GERD Evaluated by Frequency Scale for the Symptoms of GERD (FSSG) | 4 weeks
  Unit scale 0-48 was applied for an outcome measurement of the frequency of symptoms. The unit scale 0 was no symptom and scale 48 was usual symptom of GERD. The changing of the frequency of symptoms was the changing of the unit scale before and after treatment. PPI-PR GERD is defined when the changing of frequency of symptom in SSc related GERD evaluated by FSSG is improvement less than 50% compare to baseline.

SECONDARY OUTCOMES:
The proportion of participant with diffuse cutaneous SSc (dcSSc) subset between the patient who response to omeprazole and partial response to omeprazole, | 4 weeks
  The number of dcSSc subset in the patient who response to omeprazole and partial response to omeprazole, DcSSc is defined as yes or no when the patient has skin tightness includes trunk and both extremities and not include trunk and extremities, respectively.
The proportion of participant with esophageal dysphagia between the patient who response to omeprazole and partial response to omeprazole, | 4 weeks
  The number of dysphagia in the patients who response to omeprazole and partial response to omeprazole. Esophageal dysphagia is defined as yes or no when the patients has dysphagia and no dysphagia symptom, respectively.
The proportion of participant with female gender between the patient who response to omeprazole and partial response to omeprazole | 4 weeks
  The number of female gender in the patients who response to omeprazole and partial response to omeprazole. Female gender is defined as yes or no when the patient is female and male, respectively.
The proportion of participant with age>60 years between the patient who response to omeprazole and partial response to omeprazole | 4 weeks
  The number of age>60 years in the patients who response to omeprazole and partial response to omeprazole. Age>60 is defined as yes or no when the patient has age>60 and equal or less than 60 years, respectively.
The proportion of participant with modified Rodnan skin score (mRSS)>20 between the patient who response to omeprazole and partial response to omeprazole | 4 weeks
  The number of mRSS>20 in the patients who response to omeprazole and partial response to omeprazole. The mRSS was assessed at 17 sites; viz., the face, chest, abdomen, arms, forearms, hands, fingers, thighs, legs and feet. Assessment was rated as 0 (normal skin thickness), 1 (mild but definite skin thickness), 2 (moderate thickness), or 3 (sever thickness with inability to pinch a fold of skin). The score was calculated by summing the rating score from all 17 areas (range, 0-51). mRSS> 20 is defined as yes or no when the patient has mRSS>20 and equal or less than 20, respectively.
The proportion of participant with serum anti-topoisomerase I antibody positive between the patient who response to omeprazole and partial response to omeprazole | 4 weeks
  The number of anti-topoisomerase I positive in the patients who response to omeprazole and partial response to omeprazole. Serum anti-topoisomerase I antibody is defined as yes or no when the antibody in serum was positive and negative, respectively.

IPD SHARING:
Plan to Share IPD: Undecided